CLINICAL TRIAL: NCT00885469
Title: Evaluation of PillCam® ESO 2 in Patients With Suspected Esophageal Pathologies
Brief Title: PillCam® ESO 2 in Esophageal Pathologies
Acronym: MA-76
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Hila Debby -Corporate Clinical Trials Manager, Given Imaging Ltd.
Other Study IDs: MA-76
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2009-08

CONDITIONS: Barrett's Esophagus; Gastroesophageal Reflux Disease
Keywords: known Barrett's Esophagus; Suspected Barrett's Esophagus; chronic GERD; known Barrett's Esophagus or chronic GERD
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with known Barrett's Esophagus or chronic GERD

SUMMARY:
Study Hypothesis:

* PillCam™ ESO-2 will demonstrate equivalent accuracy parameters as compared to blinded esophagogastroduodenoscopy (EGD) in detecting suspected Barrett's esophagus, detecting and grading esophagitis.
* PillCam™ ESO will demonstrate all safety parameters as compared to EGD
* PillCam™ ESO-2 will demonstrate better patient's satisfaction as compared to EGD

DETAILED DESCRIPTION:
Upper endoscopy (EGD) is employed to diagnose BE; however, the cost and invasiveness of this diagnostic tool limits its utilization in many patients (17). There is a need for an alternative, simple, and less invasive diagnostic tool for evaluating GERD patients and screening for BE. Esophageal capsule endoscopy (ECE) is a novel technique that offers non-invasive evaluation of esophageal pathology in gastroesophageal reflux disease (GERD) patients. The potential benefits of screening patients by Capsule Endoscopy (CE) are several. Detection of esophageal pathology during CE could select a subgroup of patients for upper endoscopy avoiding the risks and costs of an upper endoscopy in the majority. Other benefits include convenience, ability to perform the test on an outpatient basis in less than 30 minutes, patient acceptability, minimal loss of work time, safety, tolerability, the ability of non-physicians to screen patients, and potentially, improved compliance with screening recommendations. Recently, a new, high resolution capsule (ESO 2) with a larger field of view and better illumination than the previous CE has been introduced. A simplified ingestion protocol for CE that improves visualization of the Z-line has also been reported as well (17).

ELIGIBILITY:
Inclusion Criteria:

* Patient age is 18 years or older
* Patient is known or suspected to suffer from an esophageal disease based on his/her medical history and recent symptoms suggestive of GERD or BE
* Patient agrees and signs the Informed Consent Form
* Currently taking PPI for at least 28 days.

Exclusion Criteria:

* Patient has dysphagia
* Patient has known Zenker's Diverticulum
* Patient is known or is suspected to suffer from esophageal and/or intestinal obstruction
* Patient has a cardiac pacemakers or other implanted electro medical devices
* Patient who has undergone an EGD within past seven days
* Female patient is pregnant and/or lactating
* Patient is expected to undergo Magnetic Resonance Imaging (MRI) examination within 7 days after ingestion of the capsule
* Patient has had a prior pelvic or abdominal surgery of the gastrointestinal tract (other than uncomplicated procedures that would be unlikely to lead to bowel obstruction based on the clinical judgment of the investigator such as appendectomy or uncomplicated cholecystectomy)
* Patient has any condition which precludes compliance with the study and/or device instructions
* Patient suffers from life threatening conditions
* Patient is currently participating in another clinical study
* Patient is on medications that may coat the esophagus such as iron or sulcrafate.
* Contraindication for any radiation or barium (e.g., sensitivity or allergy) required to confirm excretion of the capsule if necessary.
* Patient is currently suffering from conditions like allergy, illness (flu) or anything else that causes congestion, excessive salivation, etc. that could foster difficulty in swallowing the capsule or affect the clarity of the CE images.
* Contraindicated for use of laxatives, or surgery required to remove a capsule e.g., colonoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known Barrett's Esophagus or chronic GERD
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2007-12; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Accuracy parameters (sensitivity, specificity, NPV, PPV) of PillCam ESO 2 in detecting suspected Barrett's Esophagus (BE) as compared to standard EGD, using unblinded EGD as the reference standard. | 7 days

SECONDARY OUTCOMES:
Level of agreement (i.e. positive, negative and overall agreement parameters) between PillCam ESO 2 and standard EGD in classifying the Z-line following the ZAP score (Wallner et. al 2002), where Grades 0&I and grades II&III will be consolidated. | 7 days
Accuracy Parameters (sensitivity, specificity, NPV, PPV) of PillCam ESO 2 in detecting Esophagitis as compared to standard EGD, using unblinded EGD as the reference standard. | 7 days
Subjects' satisfaction will be assessed by a post procedure questionnaire | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Glen Eisen, MD, Principal Investigator — Oregon Health and Science University; Prateek Sharma, MD, Principal Investigator — Department of VA Medical Affairs Medical Center of Kansas City
Locations (10):
- United States (10):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - University of Illinois at Chicago, Chicago, Illinois
  - Rockford Gastroenterolgy Assoicates, Rockford, Illinois
  - Minnesota Gastroenterology, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Department of VA Medical Affairs Medical Center of Kansas City, Kansas City, Missouri
  - New York Gastroenterology Assoicates, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Virginia Mason Medical Center, Seattle, Washington